CLINICAL TRIAL: NCT06045754
Title: An Open-Label, Phase 4 Study to Evaluate the Efficacy and Safety of Dual Targeted Therapy With Vedolizumab Intravenous (IV) and Adalimumab Subcutaneous (SC) or Vedolizumab IV and Ustekinumab IV/SC in Moderate to Severe Crohn's Disease (CD)
Brief Title: A Study of Vedolizumab Intravenous (IV) and Adalimumab or Vedolizumab and Ustekinumab in Adults With Crohn's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4051; MACS-2022-120102 (Other: Study ID); EXPLORER 2.0 (Other: Takeda)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Adalimumab; Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A, Cohort 1: Vedolizumab + Adalimumab (Experimental): Participants will receive vedolizumab IV 300 mg, at Weeks 0, 2, and 6, then every 8 weeks (Q8W) until Week 22 and adalimumab SC 160, 80, and 40 mg at Weeks 0, 2, and 4, respectively, then 40 mg every 2 weeks (Q2W) until Week 26.
  Interventions: Drug: Vedolizumab; Drug: Adalimumab
- Part A, Cohort 2: Vedolizumab + Ustekinumab (Experimental): Participants will receive vedolizumab IV 300 mg, at Weeks 0, 2, and 6, then Q8W until Week 22 and ustekinumab IV 520, 390, or 260 mg (weight-based), then SC 90 mg 8 weeks after initial IV dose, then Q8W until Week 24.
  Interventions: Drug: Vedolizumab; Drug: Ustekinumab
- Part B: Vedolizumab Monotherapy (Experimental): Participants who achieve therapeutic benefit in Part A will receive vedolizumab IV 300 mg monotherapy, Q8W from Week 30 until Week 46 and will be followed up to Week 52.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion.
  Other Names: Entyvio
Drug: Adalimumab — Adalimumab subcutaneous injection.
  Other Names: Humira
  Arms: Part A, Cohort 1: Vedolizumab + Adalimumab
Drug: Ustekinumab — Ustekinumab intravenous infusion.
  Other Names: Stelara
  Arms: Part A, Cohort 2: Vedolizumab + Ustekinumab
Drug: Ustekinumab — Ustekinumab subcutaneous injection.
  Other Names: Stelara
  Arms: Part A, Cohort 2: Vedolizumab + Ustekinumab

SUMMARY:
The main aim of this study is to learn about the effect of treatment with vedolizumab IV (vedolizumab) together with adalimumab or vedolizumab (VDZ) together with ustekinumab (UST) in adults with moderate to severe Crohn's Disease, and the effect of treatment with vedolizumab alone, after the dual targeted treatment.

The study is conducted in two parts. In Part A, participants will receive the dual targeted treatment (vedolizumab together with either adalimumab or ustekinumab). In part B, participants will receive vedolizumab only. Part B will include participants who responded to the treatment in Part A.

Each participant will be followed up for at least 26 weeks after the last dose of treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is vedolizumab. Vedolizumab is being tested to treat people with moderate to severe Crohn's disease who have experienced inadequate response, loss of response or intolerance to either one prior interleukin [IL] antagonist, and no other biologic/small molecule (Group A); one IL antagonist and either one Janus kinase inhibitor (JAKi) or one TNFi (other than adalimumab) [Group B] (Cohort 1) or one prior tumor necrosis factor inhibitor [TNFi] and no other biologic/small molecule (Group C); one TNFi and either 1 JAKi or one IL antagonist (other than UST) (Group D) (Cohort 2). The study will look at the efficacy and safety of dual targeted therapy.

The study will enroll approximately 100 participants. Participants will be assigned to one of the two treatment groups in Part A:

* Part A, Cohort 1: Vedolizumab + Adalimumab
* Part A, Cohort 2: Vedolizumab + Ustekinumab

All participants who achieve therapeutic benefit in Part A will receive vedolizumab IV 300 mg monotherapy from Week 30 until Week 46 in Part B. Participants will be followed for a further 20-week safety follow-up period to Week 72 (or 26 weeks post-last dose of study drug).

This multi-center trial will be conducted in the United States and Canada. The overall time to participate in this study is approximately 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

Part A:

1. Has a confirmed diagnosis of CD at least 3 months before screening, based on endoscopy results.
2. Has moderately to severely active CD at Screening, defined as an SES-CD >=6 (>=4 if isolated ileal disease).
3. Has demonstrated at least 1 of the following (a, b, or c) to at least 1 IL antagonist or at least 1 tumor necrosis factor (TNF) antagonist, at doses approved for the treatment of CD:

   1. Inadequate response after completing the full induction regimen;
   2. Loss of response (recurrence of symptoms during scheduled maintenance dosing after prior clinical benefit); or
   3. Intolerance (a significant adverse event that precluded further use, including but not limited to serious infection including opportunistic infections, malignancy, infusion-related and hypersensitivity reactions including anaphylaxis, and liver injury).

   Note: Participants with an inadequate response to >2 classes of advanced therapies or >1 agent in the same class are not eligible. Participants who discontinued a third class of advanced therapy for reasons other than inadequate response may be eligible after discussion with the Medical Monitor.

   Part B:
4. In the investigator's opinion, the participant exhibits a therapeutic benefit at Week 26.

Exclusion Criteria:

1. CDAI score > 450.
2. A current diagnosis of ulcerative colitis or indeterminate colitis.
3. Clinical evidence of an abdominal abscess.
4. Known fistula (other than perianal fistula) or phlegmon.
5. Known perianal fistula with abscess.
6. Ileostomy, colostomy, or severe, or symptomatic stenosis of the intestine.
7. Previous extensive bowel resection with 2 entire segments missing, of the following: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum.
8. Short bowel syndrome.
9. Any planned surgical intervention for CD, except for seton placement for perianal fistula without abscess.
10. History or evidence of adenomatous colonic polyps that have not been removed.
11. History or evidence of colonic mucosal dysplasia.
12. Intolerance or contraindication to ileocolonoscopy.
13. Any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency infection).
14. Active or latent tuberculosis (TB), regardless of treatment history.
15. A positive test for hepatitis B virus (HBV) as defined by the presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) test.
16. A positive test for hepatitis C virus (HCV), as defined by a positive hepatitis C virus antibody (HCVAb) test and detectable HCV ribonucleic acid (RNA).
17. Received approved or investigational anti-integrin antibodies (i.e., vedolizumab, natalizumab, efalizumab, etrolizumab, abrilumab [AMG 181], anti- mucosal addressin cell adhesion molecule-1 [MAdCAM-1] antibodies, or rituximab) for the treatment of CD.
18. History of or symptoms of progressive multifocal leukoencephalopathy (PML) in the investigator's opinion. If a participant has symptoms consistent with PML, a PML checklist must be completed and submitted to the PML independent adjudication committee. If the PML IAC deems the participant to have PML, the participant is ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants With an Endoscopic Response Based on the Simple Endoscopic Score for (SES-CD) at Week 26 | At Week 26
  Endoscopic response is defined by a >=50 percent (%) reduction from baseline in the SES-CD. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Part B: Percentage of Participants With an Endoscopic Response Based on the SES-CD at Week 52 | At Week 52
  Endoscopic response is defined by a >=50 reduction from baseline in the SES-CD. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants in Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) (CDAI <150) at Week 12, Week 26, and Week 52 | At Weeks 12, 26, and 52
  Clinical remission is defined as a CDAI score of <150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit and body weight. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity. Percentage of participants in clinical remission based on CDAI at either Week 12, Week 26, or Week 52 will be reported in this outcome measure.
Percentage of Participants in Clinical Remission at Both Week 26 and Week 52 | At Weeks 26 and 52
  Clinical remission is defined as a CDAI score of ≤150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit and body weight. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity. Percentage of participants in clinical remission at both Week 26 and Week 52 will be reported in this outcome measure.
Percentage of Participants in 2-item Patient-reported Outcome Measure (PRO2) Remission at Weeks 12, 26, and 52 | At Weeks 12, 26 and 52
  Clinical remission based on PRO2 is defined as PRO2 score <=8 from baseline. The PRO2 is comprised of the stool frequency and abdominal pain components of the CDAI. The PRO-2 score is the sum of the abdominal pain and stool frequency subscores of the CDAI score. The average daily number of liquid or very soft stools and abdominal pain score (with 0 indicating no pain and 3 indicating severe pain) are weighted according to the CDAI multiplication factors (2 for stool frequency and 5 for abdominal pain). A higher score indicates more frequent stools and more severe abdominal pain.
Change in PRO2 Score from Week 26 to 52 | From Week 26 up to Week 52
  The PRO2 is comprised of the stool frequency and abdominal pain components of the CDAI. The PRO-2 score is the sum of the abdominal pain and stool frequency subscores of the CDAI score. The average daily number of liquid or very soft stools and abdominal pain score (with 0 indicating no pain and 3 indicating severe pain) are weighted according to the CDAI multiplication factors (2 for stool frequency and 5 for abdominal pain). A higher score indicates more frequent stools and more severe abdominal pain.
Percentage of Participants in Stool Frequency Remission | At Weeks 12, 26, and 52
  Stool frequency remission is defined as an average daily stool frequency of <=3 that is not worse than baseline.
Percentage of Participants in Abdominal Pain Remission | At Weeks 12, 26, and 52
  Abdominal pain remission is defined as an abdominal pain score of <=1 that is not worse than baseline.
Percentage of Participants in Endoscopic Remission (SES-CD 0-2) at Week 26 and Week 52 | At Weeks 26 and 52
  Endoscopic remission is defined as SES-CD score from 0-2. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease. Percentage of participants achieving endoscopic remission based on SES-CD at either Week 26 or Week 52 will be reported in this outcome measure.
Percentage of Participants in Endoscopic Remission at Both Week 26 and Week 52 | At Weeks 26 and 52
  Endoscopic remission as per SES-CD is defined as SES-CD score from 0-2. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease. Percentage of participants achieving endoscopic remission based on SES-CD at both Weeks 26 and 52 will be reported in this outcome measure.
Percentage of Participants in Deep Remission Based on the CDAI and SES-CD at Week 26 and Week 52 | At Weeks 26 and 52
  Deep remission:CDAI <150 points and SES-CD 0-2. CDAI assesses CD per clinical signs such as number of liquid/soft stools,abdominal pain,general wellbeing,extra-intestinal manifestations of CD, antidiarrheal use,presence of abdominal mass, hematocrit and body weight. It has 8 factors each summed after adjustment with weighting factor; total score:0 to 600 points, higher scores=more severity. SES-CD evaluates 4 endoscopic variables(ulcer size, percentage of ulcerated surface area, percentage of affected surface area, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0=none or not severe to 3=most severe case; sum of the scores range from 0 to 15, except for narrowing. Presence of narrowing ranges from 0 to 11. Overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables. Higher scores=more severe disease. Participants achieving deep remission at either Week 26 or 52 will be assessed in this outcome measure.
Percentage of Participants in Deep Remission at Both Week 26 and Week 52 | At Weeks 26 and Week 52
  Deep remission: CDAI <150 points and SES-CD 0-2. CDAI assesses CD per clinical signs such as number of liquid/soft stools,abdominal pain,general wellbeing,extra-intestinal manifestations of CD, antidiarrheal use,presence of abdominal mass, hematocrit and body weight. It has 8 factors each summed after adjustment with weighting factor; total score:0 to 600 points, higher scores=more severity. SES-CD evaluates 4 endoscopic variables(ulcer size, percentage of ulcerated surface area, percentage of affected surface area, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0=none or not severe to 3=most severe case; sum of the scores range from 0 to 15, except for narrowing. Presence of narrowing ranges from 0 to 11. Overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables. Higher scores=more severe disease. Participants achieving deep remission at both Weeks 26 and 52 will be assessed in this outcome measure.
Percentage of Participants With a Clinical Response (>=100-point Decrease from Baseline in CDAI Score) | At Weeks 12, 26, and 52
  Clinical response is defined as >=100-point decrease from Baseline in CDAI score. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants With Complete Endoscopic Healing | At Weeks 26 and 52
  Complete endoscopic healing is defined as SES-CD score ≤4 with a ≥2-point decrease from baseline and no individual subscore >1. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is the most severe case, with the sum of the scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Percentage of Participants Using Oral Corticosteroids at Baseline who are in Clinical Remission Based on CDAI Score and had Discontinued Corticosteroids | From Week 26 to Week 52
  Percentage of participants using oral corticosteroids at Baseline who are in clinical remission based on the CDAI score and had discontinued corticosteroids within >=30 days of Week 26 and within >= 90 days of Week 52. Clinical remission is defined as a CDAI score of ≤150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Change in SES-CD from Baseline to Week 26 and Week 52 | Baseline, Week 26 and Week 52
  SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is the most severe case, with the sum of the scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is the sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Percentage of Participants with First CD Exacerbation After 26 Weeks | From Week 26 through Week 52
  CD exacerbation is defined as a >70-point increase in CDAI from the prior visit on 2 occasions separated by a 2-week interval, and either CRP above normal or fecal calprotectin [FCP] >250 micrograms per gram (μg/g). CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Change in FCP Concentrations from Baseline to Week 12, Week 26, Week 42, and Week 52 | Baseline, Weeks 12, 26, 42, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (55):
- United States (46):
  - Digestive Health Specialsits, Dothan, Alabama
  - GI Alliance Sun City, Sun City, Arizona
  - University of California San Diego Health (UCSD), La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Clinical Research of Osceola, Kissimmee, Florida
  - Endoscopic Research Inc, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Alliance Clinical Research of Tampa, LLC, Tampa, Florida
  - Gastroenterology Consultants, P.C., Roswell, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - GI Alliance - Illinois Gastroenterology Group - Glenview, Glenview, Illinois
  - GI Alliance - Illinois Gastroenterology Group LLC - Gurnee, Gurnee, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton ONeil Clinical Research Center, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - GI Alliance, Metairie, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Huron Gastroenterology Associates, P.C., Ypsilanti, Michigan
  - Mid-America Gastro-Intestinal Consultants, Kansas City, Missouri
  - BVL Clinical Research, Liberty, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio Gastroenterology group, Inc., Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, LLC., Westlake, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network, Wexford, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - Texas Digestive Disease Consultants Cedar Park, Cedar Park, Texas
  - GI Alliance - Digestive Health Associates of Texas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Digestive Disease Consultants Lubbock, Lubbock, Texas
  - GI Alliance - Mansfield, Mansfield, Texas
  - Gastroenterology Research of San Antonio, LLC, San Antonio, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - Texas Digestive Disease Consultants (TDDC), Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - GI Alliance - Webster, Webster, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Washington Gastroenterology- GIA, Bellevue, Washington
  - Washington Gastroenterology- GIA, Tacoma, Washington
- Canada (9):
  - Covenant Health, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - West GTA Endoscopy Inc., Mississauga, Ontario
  - Viable Clinical Research - North Bay, North Bay, Ontario
  - Toronto Immune and Digestive Health Institute Inc. (TIDHI), North York, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
  - Toronto Digestive Disease Associates (TDDA) Inc., Vaughan, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/bdd5e7bc0c574c99?idFilter=%5B%22Vedolizumab-4051%22%5D